CLINICAL TRIAL: NCT07170020
Title: Hyperbaric Oxygen Treatment for Necrotizing Fasciitis and Necrotizing Soft Tissue Infections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Drue Orwig, Section Chief, Hyperbaric/Wound Care, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0980
Record Dates: First submitted 2025-08-27; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Necrotizing Fascitis
Keywords: necrotizing; fascitis; hyperbaric
MeSH Terms: conditions — Fasciitis, Necrotizing; Fasciitis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Will the hyperbaric oxygen improve morbidity and mortality compared to standard of care (Experimental): We hypothesize the addition of hyperbaric oxygen in conjunction with standard care will improve patient mortality in necrotizing soft tissue infections. This study will evaluate if the addition ofhyperbaric oxygen improves mortality in patients with necrotizing fasciitis and necrotizing soft tissue infections.
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- determine if faster diagnosis to debridement times negate the need for hyperbaric oxygen treatments (Experimental): Secondary objectives will be to evaluate the morbidity of patients treated with standard of care including hyperbaric oxygen treatments as compared to historical controls. Morbidity metrics include: decreased need for OR debridement, improved quality of life (QOL) scores, reduced mortality, reduced complications, reduced hospital length of stay.
  Interventions: Procedure: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — Hyperbaric oxygen has been shown in several case studies and retrospective studies to possibly improve mortality and morbidity in this patient population. One limitation of prior studies is many of them are retrospective. This study will be prospective.

SUMMARY:
The goal of this clinical trial is to learn if hyperbaric oxygen is beneficial in treating necrotizing infections and decreasing rates of morbidity and mortality. This study therefore has two aims:

1. Determine if hyperbaric oxygen improve morbidity and mortality compared to standard of care using a prospective model.
2. Determine if faster diagnosis to debridement times negate the need for hyperbaric oxygen treatments in necrotizing infections.

DETAILED DESCRIPTION:
Necrotizing fasciitis and necrotizing soft tissue infections are a complicated group of infections dominated largely by polymicrobial infections that rapidly spread through the skin and soft tissues. Secondary effects include vascular occlusion, ischemia, tissue necrosis, along with sepsis and multi-organ involvement. The incidence of necrotizing infections is about 6500 cases annually in the US2. There have been no major advances in disease management over the past twenty years and the mortality still ranges in the 10-43 % range2. Today early aggressive debridement and IV antibiotics remain the cornerstone of treatment. Hyperbaric oxygen has been shown in several case studies and retrospective studies to possibly improve mortality and morbidity in this patient population.1-4 One limitation of prior studies is many of them are retrospective. Additionally, not all centers are able to take patients quickly back for surgical debridement which could increase rates of morbidity and mortality. Corewell Health West Butterworth Hospital has 24/7 in-hospital acute care surgery services. This allows very short diagnosis to OR debridement wait times in necrotizing infections. This study therefore has two aims: first is to determine if hyperbaric oxygen improve morbidity and mortality compared to standard of care using a prospective model. Secondly, to determine if faster diagnosis to debridement times negate the need for hyperbaric oxygen treatments in necrotizing infections.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old
* Patients with documented necrotizing fasciitis or necrotizing soft tissue infection as assessed during initial bedside evaluation, in conjunction with available laboratory values, imaging showing gas in soft tissues consitent with necrotizing infection, or surgical debridement of necrosis of fascia, muscle, and variable levels of soft tissue involvement
* Patient or advocate is able to sign consent

Exclusion Criteria:

* Pediatric patients
* Pregnant patients
* Patients deemed unlikely to survive or unable to go to surgical debridement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-14 (Estimated); Primary Completion 2026-11-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Mortality improvement | 6 months post procedure
  To evaluate if the addition of hyperbaric oxygen improves mortality in patients with necrotizing fasciitis and necrotizing soft tissue infections.

SECONDARY OUTCOMES:
Morbitity | 6 months post procedure
  To evaluate the morbidity of patients treated with standard of care including hyperbaric oxygen treatments as compared to historical controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Corewell Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided